CLINICAL TRIAL: NCT01932255
Title: CSF Leak Following Microvascular Decompression: the Benefit of Routine Postoperative Lumbar Tap
Status: Withdrawn | Type: Observational
Why Stopped: inadequate data
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Karolinska University Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/883
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Cranial Nerve Diseases; Facial Neuralgia; Trigeminal Neuralgia; Hemifacial Spasm
Keywords: microvascular decompression surgery; cerebrospinal fluid leakage; postoperative complications
MeSH Terms: conditions — Cranial Nerve Diseases; Facial Neuralgia; Trigeminal Neuralgia; Hemifacial Spasm; Cerebrospinal Fluid Leak; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- prophylactic spinal tap: Microvascular decompression surgery approach at the Karolinska University Hospital, i.e. a small craniectomy (removal of bone without putting it back), and postoperatively serial prophylactic lumbar tap
  Interventions: Procedure: prophylactic spinal tap
- no prophylactic spinal tap: Microvascular decompression surgery approach at St Olavs Hospital Trondheim University Hospital and the University Hospital of North Norway, i.e. not comprising a policy of preventing CSF leak by performing prophylactic lumbar taps or its equivalents
  Interventions: Procedure: no prophylactic spinal tap

INTERVENTIONS:
Procedure: prophylactic spinal tap
  Groups: prophylactic spinal tap
Procedure: no prophylactic spinal tap
  Groups: no prophylactic spinal tap

SUMMARY:
Even at centers with very large experience, the risk of cerebrospinal fluid (CSF) leakage in surgery for microvascular decompression is reported up to 3%.

Prevention of leakage is important since meningitis may follow. Also, leakage usually means longer hospital stay and increased cost.

In case of detected leakage extra sutures may be applied, placement of a lumbar drain may be considered or a revision and improved closure may be attempted. With leakage in the subcutaneous tissue, but not through the skin, a local accumulation causing local symptoms may also occur. In addition to being burdensome and being associated with longer hospital stays with possible revision surgery, such complications are also very costly. The best way to reduce cost and burden, and to improve patient care, is to prevent CSF leakage.

The aim of this study is to determine if prophylactic lumbar tap is beneficial for prevention of cerebrospinal fluid leakage following microvascular decompression, by comparison of surgical approaches in 3 geographical areas in the Scandinavian health system.

Hypothesis: There is no difference in cerebrospinal fluid leakage between the group subject to prophylactic spinal tap versus the group without prophylactic spinal tap.

ELIGIBILITY:
Inclusion Criteria:

* microvascular decompression surgery for neurovascular conflict (hemifacial spasm, trigeminal neuralgia)
* surgery between 1990 and 2013
* Follow-up visit registered in medical charts > 30 days postoperatively (at either local hospital, treating neurologist or at neurosurgical clinic)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The planned study is a retrospective review of medical charts in consecutive patients undergoing surgery for neurovascular conflict by microvascular decompression surgery. Patients will be identified from the operating protocols at the respective hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
cerebrospinal fluid leakage | 30 days
  Any leakage after 3rd postoperative day (since one hospital introduces iatrogenic leakage the first 3 days after surgery)

SECONDARY OUTCOMES:
overall complication risk | 30 days
Specific complication risk | 30 days
  risks associated with prophylactic treatment: meningitis, positional head-ache (need for epidural blood-patch)
days in hospital | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Asgeir S Jakola, MD PhD, Study Chair — St. Olavs Hospital